CLINICAL TRIAL: NCT02048020
Title: Phase II Trial Of Induction Chemotherapy Followed By Attenuated Chemoradiotherapy For Locally Advanced Head And Neck Squamous Cell Carcinoma Associated With Human Papillomavirus (HPV)
Brief Title: Paclitaxel and Carboplatin Before Radiation Therapy With Paclitaxel in Treating HPV-Positive Patients With Stage III-IV Oropharynx, Hypopharynx, or Larynx Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-000915; NCI-2013-02394 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 13-000915 (Other: Jonsson Comprehensive Cancer Center); P30CA016042 (NIH)
Record Dates: First submitted 2014-01-27; First posted 2014-01-29 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Human Papilloma Virus Infection; Stage III Squamous Cell Carcinoma of the Hypopharynx; Stage III Squamous Cell Carcinoma of the Larynx; Stage III Squamous Cell Carcinoma of the Oropharynx; Stage III Verrucous Carcinoma of the Larynx; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Verrucous Carcinoma of the Larynx; Stage IVA Squamous Cell Carcinoma of the Larynx; Stage IVA Squamous Cell Carcinoma of the Oropharynx; Stage IVA Verrucous Carcinoma of the Larynx; Stage IVB Squamous Cell Carcinoma of the Larynx; Stage IVB Squamous Cell Carcinoma of the Oropharynx; Stage IVB Verrucous Carcinoma of the Larynx; Stage IVC Squamous Cell Carcinoma of the Larynx; Stage IVC Squamous Cell Carcinoma of the Oropharynx; Stage IVC Verrucous Carcinoma of the Larynx
MeSH Terms: conditions — Papillomavirus Infections; Squamous Cell Carcinoma of Head and Neck | interventions — Paclitaxel; Taxes; Carboplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (paclitaxel, carboplatin, IMRT) (Experimental): INDUCTION: Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes. Treatment repeats every 21 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.
  CHEMORADIOTHERAPY: At least 2 weeks after completion of induction chemotherapy, patients receive paclitaxel IV over 1 hour weekly and undergo IMRT daily 5 days a week for 5.5 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: paclitaxel; Drug: carboplatin; Radiation: intensity-modulated radiation therapy; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Radiation: intensity-modulated radiation therapy — Undergo IMRT
  Other Names: IMRT
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This phase II trial studies how well paclitaxel and carboplatin before radiation therapy with paclitaxel works in treating human papillomavirus (HPV)-positive patients with stage III-IV oropharynx, hypopharynx, or larynx cancer. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high energy x rays to kill tumor cells. Giving paclitaxel and carboplatin before radiation therapy with paclitaxel may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the progression-free survival at 2 years in patients with HPV-positive head and neck squamous cell carcinoma (HNSCC) who receive induction chemotherapy followed by dose de-intensified chemoradiotherapy.

SECONDARY OBJECTIVES:

I. To determine the overall survival and local-regional control for patients with HPV-positive HNSCC who receive induction chemotherapy and dose de-intensified chemoradiotherapy.

II. To determine the incidence of acute grade 3+ mucosal and esophageal toxicity associated with attenuated concurrent chemoradiotherapy in patients with HPV-positive HNSCC.

III. To determine the incidence of late toxicity in patients with HPV-positive HNSCC who receive the dose de-intensified chemoradiotherapy.

IV. To estimate the incidence of all toxicity (hematologic and non-hematologic) associated with protocol treatment for all patients on trial.

V. To estimate the response rate of HPV-positive to induction chemotherapy using carboplatin and paclitaxel.

VI. To determine the effect of reduced radiation dose on short-term and long-term quality of life among patients treated by chemoradiotherapy.

OUTLINE:

INDUCTION: Patients receive paclitaxel intravenously (IV) over 3 hours and carboplatin IV over 30 minutes. Treatment repeats every 21 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.

CHEMORADIOTHERAPY: At least 2 weeks after completion of induction chemotherapy, patients receive paclitaxel IV over 1 hour weekly and undergo intensity-modulated radiation therapy (IMRT) daily 5 days a week for 5.5 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 6, 9, and 12 months, every 3 months for 1 year, and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven (from primary lesion and/or lymph nodes) diagnosis of HPV-positive squamous cell carcinoma of the oropharynx, hypopharynx, or larynx; HPV-positivity will be defined as tumors that are p16-positive by immunohistochemistry
* Clinical stage III or IV disease; note: patients with M1 tumors are not eligible
* Appropriate stage for protocol entry, including no distant metastases, based upon the following minimum diagnostic workup:

  * History/physical examination within 4 weeks prior to registration, including assessment of weight loss in past 6 months
  * Chest x-ray (or chest computed tomography [CT] scan or positron emission tomography [PET]/CT scan) within 6 weeks prior to registration
* CT scan or magnetic resonance imaging (MRI) of the head and neck (of the primary tumor and neck nodes) and PET/CT scan
* Zubrod performance status 0-1
* Absolute neutrophil count (ANC) > 1,800 cells/mm^3
* Platelets > 100,000 cells/mm^3
* Hemoglobin (Hgb) > 8.0 g/dl (note: the use of transfusion or other intervention to achieve Hgb > 8.0 g/dl is acceptable)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 2x the upper limit of normal
* Serum creatinine =< 1.5 mg/dl or institutional upper limit of normal
* Creatinine clearance (CC) >= 50 ml/min determined by 24-hour collection or estimated by Cockcroft-Gault formula
* Negative serum pregnancy test within 7 days prior to start of induction chemotherapy (ICT) for women of childbearing potential
* Women of childbearing potential and male participants are counseled on birth control and must agree to use a medically effective means of birth control throughout their participation in the treatment phase of the study (until at least 60 days following the last study treatment)
* Patient must sign study specific informed consent prior to study entry

Exclusion Criteria:

* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years
* Patients with simultaneous primaries or bilateral tumors are excluded
* Patients who have had initial surgical treatment other than the diagnostic biopsy of the primary site or nodal sampling of the neck disease are excluded
* Patients with unknown primary tumor sites are excluded
* Patients who present with a cervical lymph node metastasis of unknown primary origin
* Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable
* Prior radiotherapy that would result in overlap of radiation therapy fields
* Primary site of tumor of oral cavity, nasopharynx, nasal cavity, paranasal sinuses, or salivary glands
* Recurrent head and neck cancer
* Current uncontrolled cardiac disease; i.e., uncontrolled hypertension, unstable angina, recent myocardial infarction (within prior 6 months), uncontrolled congestive heart failure, and cardiomyopathy with decreased ejection fraction
* Congestive heart failure with left ventricular ejection fraction < 20%
* Transmural myocardial infarction within the last 6 months
* Acute bacterial or fungal infection requiring intravenous antibiotics at registration
* Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
* Active lupus erythematosus or scleroderma with ongoing physical manifestations
* Any uncontrolled condition, which in the opinion of the investigator, would interfere in the safe and timely completion of study procedures
* Pregnant or lactating women or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception
* Prior allergic reaction to the study drug(s) involved in this protocol
* Patient is enrolled in another investigational trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-12-26 (Actual); Primary Completion 2017-01-09 (Actual); Study Completion 2017-01-09 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | From date of registration to date of first documentation of progression and/or distant metastasis, or death due to any cause, assessed at 2 years
  The true 2-year progression-free survival rate will be estimated by the proportion of efficacy-evaluable patients on study without documentation of disease progression or death 2 years from registration. A 95% confidence interval (CI) for the true progression-free survival rate will be constructed using the Duffy-Santner approach. However, Kaplan-Meier methodology will be used to estimate the final 2-year progression-free survival rate and its 95% CI in case there are censored patients.

SECONDARY OUTCOMES:
Overall survival | The time from registration to death, assessed up to 5 years
  Time to event distributions will be estimated using the Kaplan-Meier method.
Local-regional control | 2 years
  The 2-year rates of local-regional control will be calculated along with 95% CI for HPV-positive patients receiving the dose de-intensified therapy. It will also be compared with the rate from historical controls using a one-sided Z-test.
Incidence of mucosal and esophageal >= grade 3 toxicity graded according to the National Cancer Institute Common Terminology for Adverse Events version 4.0 (NCI CTCAE v4.0) | Up to 12 weeks after chemoradiotherapy
  Rates and 95% CIs of grade 3+ mucosal and esophageal toxicity, late toxicity, other toxicities, protocol treatment delivery (PTD) and death during or within 30 days of discontinuation of protocol treatment will be calculated for the patients receiving the dose de-intensified therapy.
Incidence of other >= grade 3 toxicity graded according to NCI CTCAE v4.0 | Up to 12 weeks after chemoradiotherapy
  Rates and 95% CIs of grade 3+ mucosal and esophageal toxicity, late toxicity, other toxicities, PTD and death during or within 30 days of discontinuation of protocol treatment will be calculated for the patients receiving the dose de-intensified therapy.
PTD | Up to 5 years
  Rates and 95% CIs of grade 3+ mucosal and esophageal toxicity, late toxicity, other toxicities, PTD and death during or within 30 days of discontinuation of protocol treatment will be calculated for the patients receiving the dose de-intensified therapy.
Incidence of death | During or within 30 days of discontinuation of protocol treatment
  Rates and 95% CIs of grade 3+ mucosal and esophageal toxicity, late toxicity, other toxicities, PTD and death during or within 30 days of discontinuation of protocol treatment will be calculated for the patients receiving the dose de-intensified therapy.
Quality of life as assessed by Functional Assessment of Cancer Therapy-Head & Neck (FACT-H&N) and University of Washington Quality of Life (UWQol) | Up to 5 years
  Descriptive statistics for quality of life measurements will also be obtained, using mean and standard deviation for continuous measures and frequency tables for categorical measures.

CONTACTS AND LOCATIONS:
Overall Officials: Allen Chen, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Chen AM, Felix C, Wang PC, Hsu S, Basehart V, Garst J, Beron P, Wong D, Rosove MH, Rao S, Melanson H, Kim E, Palmer D, Qi L, Kelly K, Steinberg ML, Kupelian PA, Daly ME. Reduced-dose radiotherapy for human papillomavirus-associated squamous-cell carcinoma of the oropharynx: a single-arm, phase 2 study. Lancet Oncol. 2017 Jun;18(6):803-811. doi: 10.1016/S1470-2045(17)30246-2. Epub 2017 Apr 20. PMID 28434660